CLINICAL TRIAL: NCT07064356
Title: AI-Powered Neonatal Risk Assessment for Improved Perinatal Outcomes
Status: Not yet recruiting | Type: Observational
Sponsor: FetalFirst Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: FF-NN-AI-001; IRAS ID: 358793 (Other: Health Research Authority (HRA) - Wales REC)
Record Dates: First submitted 2025-06-26; First posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Congenital Anomalies; Neonatal Complications; Perinatal Outcomes; Perinatal Outcomes of the Mother and Fetus
Keywords: Artificial Intelligence; Predictive Diagnostics; Machine Learning; Fetal Medicine; Neonatal Risk Assessment
MeSH Terms: conditions — Congenital Abnormalities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Retrospective Neonatal Data Cohort: This cohort consists of retrospective, anonymized neonatal health records, including ultrasound, MRI scans, and clinical documentation from previous cases, used to develop predictive AI models.

SUMMARY:
This study aims to develop advanced artificial intelligence (AI) models that predict neonatal risks and complications based on historical multimodal health data, including ultrasound and MRI scans. The objective is to empower clinicians and provide clear, compassionate support for families navigating complex prenatal diagnoses.

DETAILED DESCRIPTION:
The FetalFirst study employs observational, retrospective analysis utilizing DenseNet121 neural networks. It analyzes de-identified retrospective data comprising ultrasound images, MRI scans, and clinical documentation from existing medical records. This research has received ethical approval from Wales Research Ethics Committee (REC ref: 25/WA/0168, IRAS ID: 358793). Outcomes from this study are expected to significantly enhance clinical intervention strategies, offering healthcare professionals robust tools for earlier detection and improved management of congenital anomalies and neonatal risks. Additionally, the insights gained will provide critical support to parents facing high-risk pregnancies, assisting them in making informed decisions.

ELIGIBILITY:
Inclusion Criteria:

* Historical, de-identified neonatal records including ultrasound images, MRI scans, and clinical documentation available for analysis.

Exclusion Criteria:

* Cases with incomplete or missing critical data elements required for AI model analysis.

Ages: 1 Year to 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The population includes retrospective, anonymized neonatal records obtained from clinical datasets, focusing on neonates previously diagnosed or assessed for congenital anomalies and neonatal risks.
Sampling Method: Non-Probability Sample
Enrollment: 50000 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Accuracy of AI Model Predictions for Neonatal Risk | 12 Months
  Evaluate the accuracy of DenseNet121-based AI models in predicting neonatal risks and congenital anomalies, measured by sensitivity, specificity, and overall prediction accuracy.

CONTACTS AND LOCATIONS:
Overall Officials: Nawal (Nina) Abide, EMBA, MA, BA, Principal Investigator — FetalFirst Limited

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to ethical and privacy considerations. All data is pseudonymised and governed strictly by the approved Data Sharing Agreement, which restricts external sharing to protect participant confidentiality and comply with UK GDPR.

REFERENCES:
- See also: FetalFirst Project Website — https://www.fetalfirst.com